CLINICAL TRIAL: NCT06259669
Title: A US-Prospective, Registry-Based, Observational, Exposure Cohort Study to Compare Maternal, Fetal, and Infant Outcomes of Women With Mild to Moderate Atopic Dermatitis Exposed to Ruxolitinib Cream During Pregnancy With an Unexposed Control Population
Brief Title: Study to Compare Maternal, Fetal, and Infant Outcomes of Women With Mild to Moderate Atopic Dermatitis Exposed to Ruxolitinib Cream During Pregnancy With an Unexposed Control Population
Acronym: OPERA-1
Status: Recruiting | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB18424-MA-IAI-402
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Atopic Dermatitis
Keywords: ruxolitinib; Atopic Dermatitis; pruritus; eczema; topical therapy; JAK inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants of women exposed to ruxolitinib cream during pregnancy
  Interventions: Drug: Ruxolitinib Cream
- Infants of women not exposed to ruxolitinib cream during pregnancy
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib Cream
  Other Names: Opzelura

SUMMARY:
This observational (enrollment into the registry while the pregnancy is ongoing) study is being conducted to compare the frequency of major congenital malformation (MCM)s among infants of women exposed to ruxolitinib cream during pregnancy with infants of women not exposed to ruxolitinib cream during pregnancy.

DETAILED DESCRIPTION:
This study is an exposure cohort study of women within the US with AD who were exposed to ruxolitinib cream at any time during their pregnancy period, defined as up to 24 days prior to the estimated date of conception (DOC) through the end of pregnancy, compared with women in the US with Atopic Dermatitis (AD) not exposed to ruxolitinib cream during pregnancy. The DOC is estimated to occur 14 days after the last menstrual period (LMP). Eligible pregnant women may self-enroll or voluntarily be enrolled by their health care provider (HCP) by calling Syneos Health. Enrollment should occur as early in pregnancy as possible.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 15 to 50 years, with confirmed diagnosis of mild to moderate AD.
* Ability to comprehend and willingness to give informed consent for the study; a legal minor needs parental or legally authorized representative's consent.
* Prospective enrollment (ie, enrollment into the registry while the pregnancy is ongoing) or retrospective enrollment (ie, enrollment into the registry within 12 months of pregnancy outcome).
* Information available to confirm eligibility for either the exposed to ruxolitinib cream cohort or the not exposed to ruxolitinib cream cohort.

  * Ruxolitinib cream cohort: consisting of pregnancies in women with AD and exposure to at least 1 application of ruxolitinib cream during the pregnancy period.
  * Nonexposed cohort: consisting of pregnancies in women with AD but not exposed to ruxolitinib cream during the pregnancy period
* Reporter (eg, participant, maternal HCP) contact information available to allow for follow-up.
* Permission to contact the participant's and her infant's HCPs.

Exclusion Criteria:

* If no longer pregnant and pregnancy outcome occurred more than 12 months prior to enrollment.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before enrollment with another investigational medication or current enrollment in another investigational drug study.
* Any pregnancy that is exposed to any other JAK inhibitor from 5 half-lives for the specific JAK inhibitor used from LMP through the end of the first trimester for MCMs or end of pregnancy for other outcomes.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Exposure cohort study of women within the US with atopic dermatitis (AD) who were exposed to ruxolitinib cream at any time during their pregnancy period.
Sampling Method: Non-Probability Sample
Enrollment: 958 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2032-08-01 (Estimated); Study Completion 2033-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of major congenital malformation (MCM)s | Up to 12 months after birth
  Defined as any major structural or chromosomal defect in live-born infants, stillbirths or spontaneous losses equal to or greater than 20 weeks' gestation, or electively terminated pregnancies of any gestational age.

SECONDARY OUTCOMES:
Number of minor congenital malformations | Up to 12 months after birth
  Defined as abnormalities that do not significantly affect health and development, and normal variants are ascertained only among those who also have a major defect.
Number of Pregnancy outcomes | Up to birth
  Number of live births, still births, recognized spontaneous abortions and number of elective terminations as defined in the protocol.
Adverse pregnancy outcomes | Up to birth
  Number of preterm births and maternal pregnancy complications as defined in the protocol.
Gestational Age | At time of delivery
  Infant Gestational Age at birth as recorded in medical records.
Infant Sex | At time of delivery
  Infant Sex at birth as recorded in the medical records.
Infant Body Weight | At time of delivery
  Infant Body Weight at birth as recorded in medical records.
Infant Body Length | At time of delivery
  Infant Body Length at birth as recorded in medical records.
Infant Head Circumference | At time of delivery
  Infant Head Circumference at birth as recorded in medical records.
APGAR Score | At time of delivery
  One and five minute APGAR Scores at birth as recorded in medical records.
Number of small for gestational age (SGA)s | At time of delivery
  Defined as a birthweight at or below the 10th percentile for a given gestational age.
Infant Body Length | Through 12 months after birth
  Infant Body Length as recorded in medical records.
Infant Body Weight | Through 12 months after birth
  Infant Body Weight as recorded in medical records.
Infant Head Circumference | Through 12 months after birth
  Infant Head Circumference as recorded in medical records.
Abnormal development | Through 12 months after birth
  Based on Centers for Disease Control and Prevention (CDC) developmental milestones.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health (remote site), Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study to Compare Maternal, Fetal, and Infant Outcomes of Women With Mild to Moderate Atopic Dermatitis Exposed to Ruxolitinib Cream During Pregnancy With an Unexposed Control Population (OPERA-1) — https://incyteclinicaltrials.com/studies/incb18424-ma-iai-402